CLINICAL TRIAL: NCT05835882
Title: Blood Salvage From Liver Donors: a Feasibility Pilot Study. (BLEED Study)
Brief Title: Blood Salvage From Liver Donors: a Feasibility Pilot Study
Acronym: BLEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ID5429
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Liver Transplantation; Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver transplant recipients receiving blood donors' transfusion (Experimental): Liver transplant recipients in which donor blood was collected and intraoperatively transfused to recipients.
  Interventions: Biological: Red Blood Cell concentrates from organ donor

INTERVENTIONS:
Biological: Red Blood Cell concentrates from organ donor — Intervention is a 3-step procedure consisting of 1) recovering blood from the donor during organ procurement; 2) processing donor blood to RBC units; 3) transfusing donor blood to recipients, if necessary during surgery.
  1. Donor blood recovery. A: Donor evaluation. During the donor workup, the donor coordinator team gathers additional information from the donor relatives. If no contraindication to blood collection exists, the donor-recipient ABO-crossmatch is performed, and if negative the donor is considered eligible. B: Donor blood collection. It is carried out by a trained investigator, through the continuous autotransfusion system CATSmart (Fresenius Kabi) in the surgery room.
  2. Donor blood processing, carried out using the continuous flow CATSmart device. About 4 RBC units are collected.
  3. Donor RBC unit transfusion to recipients according to procedures usually adopted at our hospital (final hb level 8-9 g/dL).

SUMMARY:
Blood recovery is a common procedure that limits patient exposure to allogeneic blood products. Blood recovery is usually performed during different types of surgery, including cardiac and vascular surgery, or liver transplantation. Basically, the process utilizes blood cell savers and cell separators and is finalized to auto-transfusion. In our hospital, the blood recovery is carried out with the CATSmart continuous-flow device (Fresenius Kabi AG, Bad Homburg, Germany) that warrants the removal of > 95% of heparin, potassium, free hemoglobin, and non-emulsifiable lipids. In liver transplantation (LT), before removing the organ from the donor, the blood is usually flushed out of the liver. Nonetheless, in some circumstances, donor blood cells may be transferred to recipients together with the solid organ during graft implantation. This is a feasibility study exploring RBC (red blood cell) concentrates obtained from the blood organ donor to support transfusion requirements in liver recipients. Donor RBC units are produced according to the quality standards recommended by the European Directorate for the Quality of Medicines & HealthCare of the Council of Europe, with equivalent content of Hb and residual leukocytes as standard RBC products.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years) receiving a liver transplant from deceased donors at Fondazione Policlinico A. Gemelli IRCCS are eligible for the study.
* Liver procurement at Fondazione Policlinico A. Gemelli IRCCS.
* Identical ABO group in donor and recipient.
* Signed written informed consent to study participation.

Exclusion Criteria:

* Age <18 y.o.
* D-negative recipient with D-positive donor.
* Cytomegalovirus-negative recipient and cytomegalovirus -positive donor.
* Refusal to sign written informed consent to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number and percentage of LT recipients successfully transplanted with internal donors, who received donor RBC concentrates for the intraoperative transfusion support during liver transplant. | within surgical LT procedure
  Number and percentage of LT recipients successfully transplanted with internal donors, who received donor RBC concentrates for the intraoperative transfusion support during liver transplant.

SECONDARY OUTCOMES:
Blood product need in enrolled patients, in terms of rate of LT patients receiving no additional blood product in comparison with a control-matched series of LT patients accrued in previous observational protocol. | within surgical LT procedure
  Blood product need in enrolled patients, in terms of rate of LT patients receiving no additional blood product in comparison with a control-matched series of LT patients accrued in previous observational protocol.
Rate of graft failure in the prospective sample, as compared to controls. | 3 months
  Rate of graft failure in the prospective sample, as compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Teofili, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome, Italy